CLINICAL TRIAL: NCT06774599
Title: Effects of Nonpharmacological Interventions in Sleep Quality, Anxiety, and Delirium for Patients of Adult Intensive Care Units: a Randomized Controlled Trial
Brief Title: Effects of Nonpharmacological Interventions in Sleep Quality, Anxiety, and Delirium for Patients of Adult Intensive Care Units
Acronym: Sleep
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023079; R112-57 (Other Grant/Funding Number: Ditmanson Medical Foundation Chia-Yi Christian Hospital)
Record Dates: First submitted 2024-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Unit; Critical Care; Sleep Quality; Anxiety; Delirium
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Delirium

STUDY DESIGN:
Intervention Model Description: The experimental group (n=77, nonpharmacological intervention, and the control group (n=77, routine care). The nonpharmacological intervention involves listening of 30 mins ocean wave music, aromatherapy of lavender essential oil, and eye masks and earplugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- music combined with lavender essential oil group (Experimental): nonpharmacological intervention
  Interventions: Device: music combined with lavender essential oil group
- routine care (No Intervention): routine care

INTERVENTIONS:
Device: music combined with lavender essential oil group — listening of 30 mins ocean wave music, aromatherapy of lavender essential oil, and eye masks and earplugs.
  Arms: music combined with lavender essential oil group

SUMMARY:
This study will investigate the effect of nonpharmacological intervention in sleep quality, anxiety and delirium among adult ICU patients.

DETAILED DESCRIPTION:
Background: Due to the intensive care unit (ICU) noisy environment, nearly 66% critically ill patientsseem to suffer from poor sleep quality, which can easily lead to complications, such as anxiety, delirium, prolong hospital stay, and even increased mortality.

Objective: This study will investigate the effect of nonpharmacological intervention in sleep quality, anxiety and delirium among adult ICU patients.

Methods: The design of this study is a randomized experimental study recruiting 154 patients from five adult ICUs in a teaching hospital located in the central southern Taiwan. The experimental group (n=77, nonpharmacological intervention, and the control group (n=77, routine care). The nonpharmacological intervention involves listening of 30 mins ocean wave music, aromatherapy of lavender essential oil, and eye masks and earplugs. Research measurement tools, including demographic data, physiological index questionnaire, Richards-Campbell sleep scale (RCSQ), Chinese Visin-style sleep scale, Chinese State -Trait Anxiety Inventory-1, visual analogue scale for anxiety, which will be measured five times, before intervention (T1), every 9AM for three days (T2, T3, T4), and ICU transferring day (T5). SPSS 26.0 will be used to analyze data by using descriptive statistics, chi-square test, pearson correlation, independent t-test, paired t-test, ANOVA, generalized estimating equation (GEE).

ELIGIBILITY:
Inclusion Criteria:

* Conscious and able to speak or write (GCS ≥ 11)
* Hemodynamically stable
* Normal hearing and able to communicate in a low voice
* Stay in ICU for more than 24 hours
* Aged over 18 years.

Exclusion Criteria:

* Pre-existing insomnia diagnosis with long-term reliance on sleep medication,
* Sleep-related medical history such as sleep apnea
* Shift work prior to hospitalization
* Diagnosis of alcohol abuse or schizophrenia
* End-of-life or terminal conditions
* Allergy to essential oils
* Exclusion of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-14 (Estimated); Primary Completion 2025-10-09 (Estimated); Study Completion 2025-10-09 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality1 | To record the sleep quality at 5 times, T1: the time before treatment; T2-T4: the following three days after treatment; T5: the day leaving ICU.
  The investigator records the sleep quality using Richards-Campbell sleep scale
Sleep Quality2 | To record the sleep quality at 5 times, T1: the time before treatment; T2-T4: the following three days after treatment; T5: the day leaving ICU.
  The investigator records the sleep quality using Verran sleep scale
Anxiety1 | To record the anxiety at 5 times, T1: the time before treatment; T2-T4: the following three days after treatment; T5: the day leaving ICU.
  The investigator records the degree of anxiety using the spielberger state- trait anxiety inventory
Anxiety2 | To record the anxiety at 5 times, T1: the time before treatment; T2-T4: the following three days after treatment; T5: the day leaving ICU.
  The investigator records the degree of anxiety using the Visual analogue scale.

IPD SHARING:
Plan to Share IPD: No